CLINICAL TRIAL: NCT03405623
Title: Randomized Trial of Ultrasound-guided Radial Artery Cannulation Using Dynamic Short Axis Versus Conventional Long-axis In-plane View in Cardiac Surgery Patients.
Brief Title: Dynamic SAX vs Conventional LAX in Radial Artery Cannulation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Tae Kyong Kim, Clinical Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: DNTP vs LAX
Record Dates: First submitted 2018-01-15; First posted 2018-01-23 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Cardiac Surgical Procedures; Catheterization; Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic needle tip positioning (Active Comparator): In DNTP, SAX is used, and additionally, when the needle tip is imaged in the screen as an hyper-echoic point, the practitioner (a) moves the US probe proximally a bit, and (b) the needle is advanced until the needle tip reappears in the screen. In this manner, the practitioner repeats (a) and (b) until the needle is inserted 1 cm into the lumen of vessel, and then the catheter is inserted to finish the procedure.
  Interventions: Procedure: Dynamic needle tip positioning under ultrasound-guidance
- Conventional long-axis (Active Comparator)
  Interventions: Procedure: Conventional long-axis view

INTERVENTIONS:
Procedure: Dynamic needle tip positioning under ultrasound-guidance — The tip of needle is positioned under ultrasound-guidance using dynamic short-axis view.
  Arms: Dynamic needle tip positioning
Procedure: Conventional long-axis view — The tip of needle is positioned under ultrasound-guidance using conventional long-axis in-plane view.
  Arms: Conventional long-axis

SUMMARY:
When performing vascular cannulation such as radial artery cannulation, ultrasonography (US) helps proper positioning of the tip of needle in the vascular lumen, which facilitating cannulation of the catheter and successful pressure monitoring. Conventionally, short-axis out-of-plane (SAX) and long-axis in-plane (LAX) views are commonly used method to image the target vessel during cannulation under US guidance. Dynamic needle tip positioning (DNTP) method is newly introduced by one group of investigators who conducted a related study using vascular phantom model.

In DNTP, SAX is used, and additionally, when the needle tip is imaged in the screen as an echogenic point, the practitioner (a) proximally moves the US probe a bit, and then (b) the needle is advanced until the needle tip reappears in the screen. In this manner, the practitioner repeats (a) and (b) until the needle is inserted 1 cm into the lumen of vessel, and then the catheter is inserted to finish the procedure.

DNTP has not been compared to conventional imaging methods. The aim of this trial is to see the effect of DNTP on success rate of the radial artery cannulation at the first attempt, compared to the conventional LAX.

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiovascular surgery where RA catheterization is newly required.

Exclusion Criteria:

* skin infection or trauma
* Bilateral arteriovenous fistula for dialysis
* Severe peripheral vascular disease
* Severe arteriosclerosis or arterial atheroma
* Raynaud disease
* Shock
* Patients on ECMO or IABP support
* Morbid obesity
* Profound coagulopathy
* Negative results of modified Allen's test

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-06-04 (Actual)

PRIMARY OUTCOMES:
Success rate of the radial artery cannulation at first attempt | intraoperative
  Successful confirmation of the arterial waveform through a pressure monitor at first attempt of the radial artery cannulation

SECONDARY OUTCOMES:
Time between skin puncture to confirmation of the arterial waveform through a pressure monitoring device. | During the cannulation procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Flumignan RL, Trevisani VF, Lopes RD, Baptista-Silva JC, Flumignan CD, Nakano LC. Ultrasound guidance for arterial (other than femoral) catheterisation in adults. Cochrane Database Syst Rev. 2021 Oct 12;10(10):CD013585. doi: 10.1002/14651858.CD013585.pub2. PMID 34637140